CLINICAL TRIAL: NCT01732575
Title: Effectiveness of an Intervention Tailored for Day Centers for People With Psychiatric Disabilities
Brief Title: Enrichment of Day Centers in Community-based Psychiatry
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lund University (Other)
Collaborators: The Swedish Research Council (Other Government)
Responsible Party: Principal Investigator, Mona Eklund, Professor, Lund University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Enrich
Record Dates: First submitted 2012-11-13; First posted 2012-11-26 (Estimated); Last update posted 2015-08-25 (Estimated); Status verified 2015-08

CONDITIONS: Enrichment With Meaning-generating Activities; Rehabilitation as Usual
Keywords: everyday activities; rehabilitation; mental illness; occupational therapy
MeSH Terms: conditions — Mental Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Enrichment (Experimental): Enrichment with meaning-generating activities
  Interventions: Behavioral: Enrichment with meaning-generating activities
- Rehabilitation as usual (No Intervention): The ongoing, normal day center program.

INTERVENTIONS:
Behavioral: Enrichment with meaning-generating activities — Gaps in the rehabilitation are identified by staff and researchers in dialogue. Staff gets relevant education. An intervention is tailored by staff and researchers to bridge the gaps. Consumers have a say and the intervention is revised accordingly. The intervention is implemented and continues for 14 months.
  Arms: Enrichment

SUMMARY:
This RCT study addresses the topic of improving the possibilities for people with severe mental illness (SMI) to be engaged in meaningful daily occupations at community-based activity (CBA) centers. Meaningful occupation, which includes not only work-related activities, but also leisure, household and social activities, is assumed to generate health and wellbeing. It is well established that there is a relationship between satisfaction with daily occupations and well-being.

A Swedish mental health care reform stated that the social services should provide meaningful daily occupations to people with SMI. However, evaluations of the effects of the reform conclude that the target group's needs for meaningful daily occupation have not been met.

Thus, on the basis of governmental reports and evaluations, there is an urgent need for improving the quality of the activities and support offered at CBA centers. Therefore, the overarching aim of this project is to develop and implement an intervention method for improving the activities offered and support given at CBA centers, and evaluate the outcomes of that intervention.

Specific aims

* Developing and implementing an intervention that means reorganization of CBA centers in such a way that they become enriched with characteristics that have been identified as rewarding and meaningful in previous research.
* Evaluating the outcome of that intervention on:

  * the unit level, i.e., in terms of changes in the characteristics of the CBA centers,
  * the individual level, in terms of changes among the consumers regarding satisfaction with the activities at the CBA center, perceived control, social interaction, quality of life, etc.

Cluster randomization is used. Day centers are randomized to either giving the new intervention ("enrichment") or continuing with "care as usual" during the study period, which is 14 months. This means that all participants in a day center get the type care their specific day center offers during the study period.

ELIGIBILITY:
Inclusion Criteria:

* severe mental illness > 2 years
* age 18-65 years
* visiting the day center > 4 hrs per week

Exclusion Criteria:

* comorbidity of dementia or developmental disorder
* acute psychosis
* primary diagnosis of substance use disorder
* insufficient knowledge of Swedish

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2008-10; Primary Completion 2012-02 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Score on questionnaire regarding perceived meaning in day center occupations | Up to 14 months
  A self-report measure, Estimation of Perceived Meaning in Day Centers (EPM-DC,) has been developed in previous research. It is a psychometrically sound instrument for assessing meaningfulness in the day center context.
  Nilsson, I., Argentzell, E., Sandlund, M., Leufstadius, C., & Eklund, M. (2011). Measuring perceived meaningfulness in day centres for persons with mental illness. Scand J Occup Ther, 18(4), 312-320.

SECONDARY OUTCOMES:
Score on satisfction with the rehabilitation | Up to 14 months
  The instrument is widely used an well-tested. It is a self-report measure that targets satisfaction with the care/rehabilitation received.
  Larsen, D. L., Attkisson, C. C., Hargreaves, W. A., & Nguyen, T. D. (1979). Assessment of client/patient satisfaction: development of a general scale. Eval Program Plann, 2(3), 197-207.

OTHER OUTCOMES:
Quality of life score | Up to 14 monts
  The individual assesses his/her quality of life according to the MANSA scale, which is a self-report measure asking for satisfaction in 11 life domains.
  Priebe, S., Huxley, P., Knight, S., & Evans, S. (1999). Application and results of the Manchester Short Assessment of Quality of Life (MANSA). Int J Soc Psychiatry, 45(1), 7-12.

REFERENCES:
- [Derived] Eklund M, Sandlund M. Predictors of valued everyday occupations, empowerment and satisfaction in day centres: implications for services for persons with psychiatric disabilities. Scand J Caring Sci. 2014 Sep;28(3):582-90. doi: 10.1111/scs.12085. Epub 2013 Oct 8. PMID 25066326